CLINICAL TRIAL: NCT04489550
Title: Optimal Duration of Magnetic Resonance Imaging (MRI) Follow-up to Safely Identify Middle Ear Residual Cholesteatoma
Brief Title: How Long Must the MRI Follow-up Last to Safely Identify Middle Ear Residual Cholesteatoma
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0224
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Middle Ear Cholesteatoma
Keywords: residual cholesteatoma; imaging follow-up; canal wall-up tympanoplasty; non-EP DWI
MeSH Terms: conditions — Cholesteatoma, Middle Ear

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Previous studies demonstrated the high diagnostic value of non-echoplanar diffusion weighted magnetic resonance imaging (non-EP DWI) for residual cholesteatoma. However, limited data are available regarding a suitable length of imaging follow-up. The present study aimed to determine the optimal duration of non-EP DWI follow-up for residual cholesteatoma

DETAILED DESCRIPTION:
A retrospective, monocentric study was performed between 2013 and 2019 and included all patients regularly followed-up after canal wall-up tympanoplasty with at least two non-EP DWI performed on the same 1.5T MRI scanner. MR images were reviewed independently by two radiologists. Sensitivity and specificity values were calculated as a function of time after the surgery. Receiver operating characteristics (ROC) curves were analyzed to determine the optimal follow-up duration.

ELIGIBILITY:
Inclusion criteria:

- patients regularly followed-up for middle ear cholesteatoma, who underwent two or more non-EP DWI performed on the same 1.5 Tesla MRI scanner

Exclusion criteria:

- congenital cholesteatomas, tympanoplasty with canal wall-down technique, or suspicion of residual cholesteatoma on the first MRI follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with history of middle-ear cholesteatoma, who underwent canal wall-up tympanoplasty and are therefore at risk of residual cholesteatoma
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
MRI sensitivity and specificity values as a function of the duration of the follow-up | 1 day
  MRI sensitivity and specificity values as a function of the duration of the follow-up. Since no official recommendations are available in the literature, the decision regarding the number of MRIs and the time lapse between any two was left to the discretion of the surgeon

SECONDARY OUTCOMES:
Receiver operating characteristics (ROC) curves | 1 day
  the receiver operating characteristics (ROC) curves

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Venail, MD, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC